CLINICAL TRIAL: NCT01112865
Title: A Multicenter, Open-label, Randomized Two Arm Cross Over Study Assessing Dyad (Subject and Caregiver) and Adult Subject Perception of Convenience and Preference of the Newly Developed Genotropin Mark VII Pen.
Brief Title: Cross Over Convenience And Preference Study Of New Mark VII Compared To Genotropin Pen In Pediatric And Adult Subjects
Acronym: CHOOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A6281297
Record Dates: First submitted 2010-04-20; First posted 2010-04-28 (Estimated); Results first posted 2012-05-14 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone Deficiency; Somatropin; Injection Pen; Medical Device; Cross Over Study; Preference; Convenience; Children; Dyads; Adults
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mark VII/Current pen (Other): Subject will use Mark VII pen for 2 months followed by Current pen for 2 months
  Interventions: Device: Genotropin Pen; Device: MARK VII pen
- Current pen/Mark VII (Other): Subject will use current Genotropin pen for 2 months followed by Mark VII pen for 2 months
  Interventions: Device: Genotropin Pen; Device: MARK VII pen

INTERVENTIONS:
Device: Genotropin Pen — Pen provided in 5, 5.3 and 12 mg doses, Dose based on body weight, subcutaneous injection daily for 2 months while in study.
  Arms: Mark VII/Current pen
Device: MARK VII pen — Pen provided in 5, 5.3 and 12mg doses, dose based on body weight, subcutaneous injection daily for 2 months while in study.
  Arms: Mark VII/Current pen
Device: Genotropin Pen — Pen provided in 5, 5.3 and 12mg doses, dose based on body weight, subcutaneous injection daily for 2 months while in study.
  Arms: Current pen/Mark VII
Device: MARK VII pen — Pen provided in 5, 5.3 and 12mg doses, dose based on body weight, subcutaneous injection daily for 2 months while in study.
  Arms: Current pen/Mark VII

SUMMARY:
Convenience and preference for the new Mark VII pen compared to the current Genotropin pen will be assessed using a questionaire. it is expected that the new pen will be preferred or at least no different to the current pen.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 8 years.
* Subjects who are starting treatment with growth hormone (Genotropin) for the first time.

Exclusion Criteria:

* Subjects with Prader-Willi syndrome or chronic renal insufficiency.
* Subjects and caregivers who, in the opinion of the investigator are not able to adequately participate in the study.
* Subjects with chronic systemic disorders, such as diabetes and heart disease.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno - Mesto
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- Germany (5):
  - Vestische Kinder- und Jugendklinik Datteln, Datteln
  - Universitaetsklinik fuer Kinder und Jugendliche, Erlangen
  - Privatpraxis, Gauting
  - Praxis fuer paediatrische Endokrinologie, Niederrad
  - Privatpraxis, Oldenburg
- Netherlands (2):
  - Sophia Kinderziekenhuis, Rotterdam
  - Juliana Kinderziekenhuis / Endocrinologie, The Hague
- Slovakia (2):
  - Narodny endokrinologicky a diabetologicky ustav, Ľubochňa, Slovakia
  - Detska fakultna nemonica s poliklinikou, II. Detska klinika, Bratislava
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Centrum for Endokrinologi och Metabolism (CEM), Gothenburg
  - Drottning Silvias barn- och ungdomssjukhus, SU/Ostra, Gothenburg
  - Barn och Ungdomsmedicinkliniken, Linköping
  - Barnmedicinkliniken N, Umeå
- Turkey (Türkiye) (2):
  - Ankara University Medical Faculty Department of Internal Diseases, Sihhiye, Ankara
  - Istanbul University Istanbul Medical Faculty Department of Pediatric Health and Diseases, Çapa, Istanbul
- United Kingdom (4):
  - Salford Royal NHS Foundation Trust, Hope Hospital, Salford, Manchester
  - Royal Hospital for Sick Children, Glasgow
  - St Thomas Hospital, London
  - Norfolk and Norwich University Hospital, Norwich

REFERENCES:
- [Derived] Pleil AM, Darendeliler F, Dorr HG, Hutchinson K, Wollmann HA. Results from an international multicenter trial evaluating the ease-of-use of and preference for a newly developed disposable injection pen for the treatment of growth hormone deficiency in treatment-naive children and adults. Med Devices (Auckl). 2014 Apr 11;7:61-71. doi: 10.2147/MDER.S59821. eCollection 2014. PMID 24748824
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281297&StudyName=Cross%20Over%20Convenience%20And%20Preference%20Study%20Of%20New%20Mark%20VII%20Compared%20To%20Genotropin%20Pen%20In%20Pediatric%20And%20Adult%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Mark VII Pen Then Genotropin® Pen: Participant (not caregiver) used Mark VII pen (subcutaneous injections daily for 2 months) then the current Genotropin® pen (subcutaneous injections daily for 2 months). Both pens provided in 5, 5.3, and 12 mg doses of Genotropin (somatropin recombinant deoxyribonucleic acid [rDNA] origin); doses received by participants based on body weight.
- Genotropin® Pen Then Mark VII Pen: Participant (not caregiver) used current Genotropin® pen (subcutaneous injections daily for 2 months) then the Mark VII pen (subcutaneous injections daily 2 months). Both pens provided in 5, 5.3, and 12 mg doses of Genotropin (somatropin [rDNA origin]); doses received by participants based on body weight.
Period: First Intervention
Arm/Group | Mark VII Pen Then Genotropin® Pen | Genotropin® Pen Then Mark VII Pen
Started | 59 | 61
Completed | 59 | 61
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Mark VII Pen Then Genotropin® Pen | Genotropin® Pen Then Mark VII Pen
Started | 59 | 61
Completed | 59 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to first use the Mark VII pen (subcutaneous injections daily for 2 months) and participants randomized to first use the current Genotropin® pen (subcutaneous injections daily 2 months). Both pens provided in 5, 5.3, and 12 mg doses of Genotropin (somatropin [rDNA origin]); doses received by participants based on body weight.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 120
Age, Customized [Number; unit: participants]
  ≤7 years | 28
  Between 8 and 17 years | 50
  Between 18 and 44 years | 18
  Between 45 and 64 years | 22
  ≥65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 69

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Dyads (Participant and Caregiver or Parent) and Adult Participants Reporting no Difference or Easier to Use for the New Genotropin Mark VII Injection Pen Compared to the Genotropin Pen®
Description: Participants were asked the following question from Section II of the Injection Pen Assessment Questionnaire (IPAQ) patient-reported outcome (PRO) tool, "Thinking about the Genotropin pen and the new injection pen you used over the past few months, please compare both injection pens and choose which one is easier to use overall?" Choices included: Genotropin Pen® easier to use, new injection pen easier to use, or no difference.
Time Frame: Month 4
Population: Full Analysis Set (FAS): randomized participants who used a study pen at least once to administer somatropin; Number of participants analyzed (N)= participants with evaluable data. Dyad defined as the participant (child being treated) and adult partner (parent or caregiver).
Measure: Number (95% Confidence Interval); unit: percentage of dyads, adult participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 119
percentage of dyads, adult participants | 67.23 [58.79 to 75.66]

2. Secondary Outcome: Percentage of Dyads and Adult Participants Reporting no Preference or Preference for the New Genotropin Mark VII Injection Pen Compared to the Genotropin Pen®
Description: Participants were asked the following question from Section II of the IPAQ PRO tool, "Thinking about both injection pens over the past few months, please choose which injection pen you prefer overall." Choices included: prefer Genotropin Pen®, prefer new injection pen, or no preference.
Time Frame: Month 4
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of dyads, adult participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 120
percentage of dyads, adult participants | 64.17 [55.59 to 72.75]

3. Secondary Outcome: Percentage of Dyads and Adult Participants Reporting the New Genotropin Mark VII Injection Pen Easier to Use Compared to the Genotropin Pen®
Description: Participants were asked the following question from Section II of the IPAQ PRO tool, "Thinking about the Genotropin pen and the new injection pen you used over the past few months, please compare both injection pens and choose which one is easier to use overall?" Choices included: Genotropin Pen® easier to use, new injection pen easier to use, or no difference.
Time Frame: Month 4
Population: FAS; Number of participants analyzed (N)= participants with evaluable data
Measure: Number (95% Confidence Interval); unit: percentage of dyads, adult participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 119
percentage of dyads, adult participants | 51.26 [42.28 to 60.24]

4. Secondary Outcome: Percentage of Dyads and Adult Participants Reporting the New Genotropin Mark VII Injection Pen Preferable Compared to the Genotropin Pen®
Description: as for outcome 2
Time Frame: Month 4
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of dyads, adult participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 120
percentage of dyads, adult participants | 54.17 [45.25 to 63.08]

5. Secondary Outcome: Percentage of Dyads and Adult Participants Who Would Choose the New Genotropin Mark VII Injection Pen in Preference to the Genotropin® Pen
Description: Investigators were asked the following study treatment continuation question, "Which device did the participant choose for continued treatment?" Choices included the Genotropin® Pen or the new injection pen.
Time Frame: Month 4
Population: FAS subset of participants located in areas where the new device was available.
Measure: Number (95% Confidence Interval); unit: percentage of dyads, adult participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 55
percentage of dyads, adult participants | 47.27 [34.08 to 60.47]
Statistical Analysis 1: Comparison: Entire Study Population; Null hypothesis: percentage of participants preferring Genotropin Mark VII injection pen = 50%; Test type: Superiority or Other; p = 0.6858, binomial test — Binomial test against the null hypothesis

6. Secondary Outcome: Ease of Use of Each Injection Pen
Description: Participants were asked the following question from Section I of the IPAQ PRO tool, "Thinking about the injection pen you have been using for the past few months, how easy or difficult it is for you to use the injection pen overall?" Responses were provided using a 5 point scale which ranged from very easy (5), somewhat easy (4), neither easy nor difficult (3), somewhat difficult (2), or very difficult (1).
Time Frame: Month 2 and Month 4
Population: FAS; Number of participants analyzed (N) = participants with evaluable data
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Mark VII Pen: Participants who used the Mark VII pen (subcutaneous injections daily for 2 months) any time during the study. Pens provided in 5, 5.3, and 12 mg doses of Genotropin (somatropin recombinant deoxyribonucleic acid [rDNA] origin); doses received by participants based on body weight.
- Genotropin® Pen: Participants who used the current Genotropin® pen (subcutaneous injections daily for 2 months) anytime during the study. Pens provided in 5, 5.3, and 12 mg doses of Genotropin (somatropin [rDNA origin]); doses received by participants based on body weight.
Arm/Group | Mark VII Pen | Genotropin® Pen
Number analyzed (Participants) | 119 | 119
scores on a scale | 4.5 (0.64) | 4.2 (0.71)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Safety Population: All randomized participants who used a study pen (Genotropin® pen or the new Mark VII injection pen) at least once to administer Genotropin.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 2/120
Other Adverse Events (participants affected / at risk) | 48/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=120)
Diarrhoea (Gastrointestinal disorders) | 1
Laryngitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=120)
Ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Application site pain (General disorders) | 1
Fatigue (General disorders) | 1
Injection site haematoma (General disorders) | 2
Injection site haemorrhage (General disorders) | 1
Injection site injury (General disorders) | 4
Injection site pain (General disorders) | 4
Injection site reaction (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 7
Otitis media (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 4
Respiratory tract infection viral (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 6
Accidental overdose (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.